CLINICAL TRIAL: NCT04966728
Title: Ultrasonic Diagnosis of Tear of the Anterior Superior Labrum of the Hip
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018096
Record Dates: First submitted 2021-06-27; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Acetabular Labrum Tear

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- suspected tear of the anterior superior labrum of the hip: One group consisted of patients with suspected tear of the anterior superior labrum of the hip.
  Interventions: Diagnostic Test: conventional ultrasound diagnosis of the hip joint, contrast-enhanced ultrasound, and high-resolution single hip MRI
- non-hip joint diseases: For non-hip joint reasons, come to the ultrasound department of our hospital to diagnose patients at the same time, and exclude other past and current hip diseases
  Interventions: Diagnostic Test: conventional ultrasound diagnosis of the hip joint, contrast-enhanced ultrasound, and high-resolution single hip MRI

INTERVENTIONS:
Diagnostic Test: conventional ultrasound diagnosis of the hip joint, contrast-enhanced ultrasound, and high-resolution single hip MRI — conventional ultrasound diagnosis of the hip joint, contrast-enhanced ultrasound, and high-resolution single hip MRI

SUMMARY:
The patients were divided into two groups, one group was a suspected hip joint anterior superior labrum tear, and the other group was a non-hip joint disease. The patients received conventional ultrasound diagnosis of the hip joint, contrast-enhanced ultrasound, and high-resolution single hip MRI for surgery Perform diagnostic power test for the gold standard.

DETAILED DESCRIPTION:
The patients were divided into two groups, one group was patients with suspected anterior superior labrum tear, and the other group was patients with non-hip joint diseases. Routine ultrasound diagnosis of the hip, contrast-enhanced ultrasound, and high-resolution single hip MRI were performed. For patients undergoing hip arthroscopic surgery after diagnostic occlusive treatment, the results of arthroscopic exploration are used as the diagnostic gold standard. A tear detected during the operation was judged to be positive, and a tear not detected was judged to be negative. For patients who have not undergone hip arthroscopic surgery after the closure treatment, if the MRI of the hip is performed, the MRI result is the gold standard. The diagnosis of tearing was judged as positive, and the undiagnosed tearing was judged as negative. This study was used to compare (1) the diagnostic efficacy of hip joint contrast-enhanced ultrasound and high-resolution single hip MRI in patients with suspected anterior superior labrum tear. (2) Comparison of the diagnostic efficiency of contrast-enhanced hip joint ultrasound and conventional ultrasound in patients with suspected anterior superior labrum tear. (3) In the process of judging the hip joint anterior superior labrum tear by conventional ultrasound and contrast-enhanced ultrasound of the hip joint, the consistency of repeated readings and the comparison of the consistency between readers.

ELIGIBILITY:
Inclusion Criteria:

Case group inclusion criteria (1) Age is greater than or equal to 18 years old (2) Patients with preoperative ultrasound examination for clinically planned hip joint anterior superior labrum tear (3) The patient can understand and sign the informed consent form .

Control group inclusion criteria

1. Age is greater than or equal to 18 years old
2. Patients who come to the ultrasound department of our hospital for treatment of non-hip joints at the same time
3. The patient can understand and sign the informed consent form

Exclusion Criteria:

Case group exclusion criteria

1. Mental conditions are not allowed
2. Adhesives that are allergic to any known . Control group exclusion criteria (1) Mental conditions are not allowed (2) Adhesives that are allergic to any known (3) Past and current diseases of other hip joint diseases

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Case group: Outpatient Department of Sports Medicine, Peking University Third Hospital, clinically diagnosed patients with hip joint labrum tear, preoperative ultrasound examination. Control group: Patients who came to our hospital's ultrasound department at the same time for non-hip joint reasons matched by age, gender and case group.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Comparison of conventional ultrasound diagnosis of the hip joint and arthroscopic diagnosis results | Hip arthroscopy was performed 1 week after ultrasound diagnosis of the hip joint.
  Comparison of conventional ultrasound diagnosis of the hip joint and arthroscopic diagnosis results
Comparison of conventional contrast-enhanced ultrasound diagnosis of the hip joint and arthroscopic diagnosis results | Hip arthroscopy was performed 1 week after conventional contrast-enhanced ultrasound diagnosis of the hip joint.
  Comparison of conventional contrast-enhanced ultrasound diagnosis of the hip joint and arthroscopic diagnosis results
Comparison of high-resolution single MRI diagnosis of the hip joint and arthroscopic diagnosis results | Hip arthroscopy was performed 1 week after high-resolution single MRI diagnosis of the hip joint.
  Comparison of high-resolution single MRI diagnosis of the hip joint and arthroscopic diagnosis results

CONTACTS AND LOCATIONS:
Overall Officials: Ligang Cui, Study Chair — Peking University Third Hospital
Locations (1):
- Department of Ultrasound Diagnosis, Peking University Third Hospital, Beijing, Beijing Municipality, China